CLINICAL TRIAL: NCT06672627
Title: Trueness of Digital Occlusal Analysis Using Handheld Device Versus Intraoral Scanner (A Diagnostic Evaluative Clinical Study)
Brief Title: Trueness of Digital Occlusal Analysis
Status: Active, not recruiting | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rania Elsayed, Lecturer, Department of Prosthodontics, Alexandria University
Other Study IDs: 0974-09
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Dental Occlusion; Occlusal Analysis
Keywords: Occlusal analysis; Occlusense; Intraoral scanners
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Every participant will undergo occlusal analysis using conventional methods (8um articulating paper)
- Study group I: Every participant will undergo digital occlusal analysis using hand held device (occlusense)
- Study group II: Every participant will undergo digital occlusal analysis using intraoral scanner (Medit occlusal analyzer)

SUMMARY:
The aims of this observational study are to evaluate the trueness of two different digital occlusal analyzers; handheld occlusal analyzer versus intraoral scanner in comparison to conventional methods in identifying true occlusal contacts and to evaluate inter-examiner reliability of two examiners independently analyzing occlusal contacts.

DETAILED DESCRIPTION:
Evaluate the trueness of two different digital occlusal analyzers; handheld occlusal analyzer (occlusense) versus intraoral scanner (Medit i700-medit occlusal analyzer) in comparison to conventional methods (8 um articulating paper) in identifying true occlusal contacts and to evaluate inter-examiner reliability of two examiners independently analyzing occlusal contacts.

ELIGIBILITY:
Inclusion Criteria:

* Normal occlusion (Angle Class 1)
* No missing teeth
* No tempromandibular disorders

Exclusion Criteria:

Patients having:

* Dental prostheses
* Extensive restorations
* Severe malocclusion
* Periodontal disease
* Excessive tooth wear
* Orofacial pain
* Temporomandibular joint disorders
* Anterior or posterior open bite
* Active orthodontic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of trueness | 4 months
  Trueness is defined as the closeness of the measurement to the real size of an object. The trueness of handheld occlusal analyzers (occlusense) versus intraoral scanners (medit occlusal analyzer) will be evaluated in comparison to conventional methods (8 um articulating paper).

SECONDARY OUTCOMES:
Inter-examiner reliability | 4 months
  Two examiners will record independently the interocclusal contacts for all the different groups, classifying them in a dichotomy variable (yes/no) contact or not per tooth. Then, the inter-examiner's reliability will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Rania Elsayed Ramadan, PhD, Principal Investigator — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt